CLINICAL TRIAL: NCT03984331
Title: MariGen Fish Skin Compared to Cadaver Skin as a Temporary Covering for Full Thickness Burns: An Early Feasibility Trial
Brief Title: Fish Skin Compared to Cadaver Skin as Temporary Cover for Full Thickness Burns
Acronym: Kereburn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerecis Ltd. (Industry)
Collaborators: MedStar Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS-0340 - P2587; CDMRP-MB150220 (Other Grant/Funding Number: MBRP)
Record Dates: First submitted 2019-01-10; First posted 2019-06-13 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Burns
Keywords: Fish skin; Full thickness burn; Burns; Cadaver Skin; Split Thickness Skin Graft; Temporary Cover; Blaze; Kerecis
MeSH Terms: conditions — Burns; Ichthyosis Vulgaris

STUDY DESIGN:
Intervention Model Description: Two adjacent burn sites on the body of each burn patient will be randomized to receive initial early cover treatment after debridement with either fish skin or cadaver skin for 7± 3 days. After the initial 7± 3 days the test sites will be grafted with STSG.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The burn wound trial area consists of two adjacent burn wound sites. The randomization will happen on the day of debridement. The test areas will be randomized to treatment so that one side receives early cover with fish skin and the other one with SOC. Treating physician will be aware of which product is being used on each site as temporary cover before grafting, but will not give this information to the patient. Prior to grafting, a blinded burn surgeon investigator will assess the burn wound bed. He/she will only have a subject number. The same procedure is used for the secondary endpoints of local reactions. Reassessment done by treating physician before STSG cannot be blinded as it is obvious what temporary treatment the test areas have received. Photos taken of wounds during the treatment (where products are not visible) will be judged blind by additional investigators. Scar assessment at 3 and 12 months via the Vancouver Scar Sale will also be fully blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Fish skin (Experimental): All patients will receive both treatments, fish skin and cadaver skin, as early cover after early debridement. This group of wounds will receive only fish skin.
  Interventions: Device: Fish skin
- Cadaver skin (Active Comparator): All patients will receive both treatments, fish skin and cadaver skin, as early cover after early debridement. This group of wounds will receive only cadaver skin.
  Interventions: Device: Cadaver skin

INTERVENTIONS:
Device: Fish skin — One out of two adjacent burn sites of 10-20 cm x 7cm surface area will be randomized to receive fish skin as early cover. Each patient thus serves as his/her own control. After 7 +/- 3 days the burn site will receive a meshed split thickness skin graft.
  Other Names: Marigen TM; Kerecis Omega3 Burn
  Arms: Fish skin
Device: Cadaver skin — One out of two adjacent burn sites of 10-20 cm x 7cm surface area will be randomized to receive cadaver skin as early cover. Each patient thus serves as his/her own control. After 7 +/- 3 days the burn site will receive a meshed split thickness skin graft.
  Arms: Cadaver skin

SUMMARY:
Objectives and rationale: Optimal burn management involves removing all the dead or burned tissue as early as feasible and cover with an autograft called split thickness skin graft (STSG) taken from the patient. This procedure creates a new wound on the patient and sometimes, when the burn covers very large portion of the patient body, there is a lack of healthy skin to use for this purpose. Under those circumstances, donated cadaver skin is used as a temporary coverage until the patient´s own donor site wound has healed enough to be used again.

The proposed clinical study aims to determine if treatment with fish skin is an alternative to cadaver skin as a temporary coverage for debrided full-thickness burns prior to STSG in terms of autograft take, time to heal, quality of healing (scarring), pain and adverse effects.

DETAILED DESCRIPTION:
Mortality after severe burns has diminished during the last decades and survival is no longer considered the primary end point of care. More attention is paid to the final functional and cosmetic outcome of the affected area but outcomes are still far from optimal. For the time being, one of the main goals in burn treatment is to achieve reduced scar formation from the time of injury. A temporary or permanent covering of the wound bed should be achieved at the time of excision. In burn wounds the gold standard is to use split thickness skin graft, or STSG, which includes epidermis, basement membrane, and a part of upper dermis. Yet the use of skin grafts has many shortcomings: there is only a limited amount of skin available for grafting, the donor sites are susceptible to infections, to pain, to pigmentation changes, and to scarring especially when re harvested. Therefore, for complicated burns, initial treatment is often with temporary coverage where cadaver skin has been the accepted standard of care.

In recent years there has been progress in the development of advanced wound care products. This has resulted in a third generation of wound treatment, known as acellular dermal grafts or skin substitutes.

Aims The goal of this clinical trial is to demonstrate that fish skin is an alternative to cadaver skin as early cover before STSG in burn wounds. This trial will be open to patients who are scheduled to receive meshed STSG of any ratio. Fish skin or cadaver skin will be applied after initial debridement in order to prepare the wound area for STSG.

5 to 10 patients will be prospectively enrolled and two burn sites on their body will randomized to initial treatment after debridement with either fish skin or cadaver skin for 7+/-3 days. After the initial treatment, the test sites will be grafted with STSG.

The histological differences and the functional outcomes will be assessed for 12 months.

Products will be applied by experienced burn surgeons at a burn center. At approximately Day 7, or when the treating physician deems the wound to be ready for grafting, the products will be removed. Prior to grafting, a second blinded burn surgeon will assess the burn wound bed.

Important dates for blinding are on Day 7 prior to STSG treatment and on Days 14, 21 and 28 for graft take, epithelialisation and wound closure. Scar assessment at 3 and 12 months via the Vancouver Scar Sale will also be fully blinded.

Key interventions:

Randomized to either cadaver skin or fish skin after initial debridement Two areas each of 10-20 x 7 cm side by side. Other areas will be treated as per local Standard of care (SOC). Concomitant medications will be given, e.g. painkiller, antibiotics, as needed.

Wound dressings changed approximately every three days until allograft or xenograft removal.

Approximately one week after placement the fish skin and cadaver allografts removed as required.

Subsequent meshed autograft placement if donor sites are available. Autografts covered with secondary antimicrobial/silver dressing and dressings approximately every 3 days until healed.

Autografts monitored for adherence, color, autograft take, and visual signs of infection.

During the operation, a 3 or 4 mm punch biopsy will be harvested from the excised wound bed before covering with any material.

ELIGIBILITY:
Inclusion Criteria:

* Participant or legally authorized representative is willing and able to give informed consent for participation in the clinical trial.

  * Patients from 22 to 75 years of age. Acute full thickness burn wounds outside the following areas; facial, genital and across joints, requiring widely meshed skin grafting or staging of STSG treatment due to insufficient healthy donor sites.
  * Maximal Total Body Surface Area (TBSA) of 50% full thickness burns
  * Able (in the Investigators opinion) and willing to comply with all clinical trial requirements.
  * Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the clinical trial.

Exclusion Criteria:

* Declined consent

  * Immunocompromised patients or patients receiving immunosuppressive therapy
  * Presently participating in another clinical trial
  * Patient actively taking glucocorticoid or cytostatic medications
  * Persons with immune deficiency because of disease or iatrogenic-
  * Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the clinical trial, or may influence the result of the clinical trial, or the participant's ability to participate in the clinical trial.
  * Patient has known allergy to fish. (Shell fish allergy is not a contraindication)
  * Exclusion areas are, facial, genital and across joints.
  * Female participants who are pregnant, breast feeding or planning pregnancy during the course of the clinical trial

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Proportions of wounds that have healed | At 3 weeks days after STSG
  Wounds which have reached at least 95% epithelialization

SECONDARY OUTCOMES:
Percentage of wound area exhibiting graft failure | At 2 weeks after STSG
  The proportion of the wound area in which the graft does not take
Full epithelialization of wound | At 2 weeks after STSG
  Number of wounds fully epithelialized
Scarring estimated with the Vancouver Scar Scale (VSS) | At 12 months after STSG
  Vascularity (0-3), pigmentation (0-3), pliability (0-3), height (0-3), Total score;0=Best, 12=worst
Inflammation profiling of wound punch biopsies as assessed by histology | Before STSG, 2 and 3 weeks and 12 months after STSG
  Histological analysis of punch wound biopsies via standard H&E staining, or staining for known inflammatory markers (TNF-alpha, IL-1b, IL-6, IL-8)
Average number of antibiotics treatments per patient | At all treatments appointments until 4 weeks after STSG
  Average number of antibiotics treatments per patient
Pain assessed by the Visual Analog Scale (VAS) before and after dressing changes | At all treatments appointments until 3 weeks after STSG
  Pain by the Visual Analog Scale (VAS) on a scale of 0-10, 0=no pain, 10= pain as bad as it could be
Bleeding time | At all treatments appointments until 3 weeks after STSG
  Average time in seconds to achieve hemostasis during dressing changes
Dermatitis | At all treatments appointments until 3 weeks after STSG
  Incidence of dermatitis
Ease-of-use | Day 0 when grafts are initially applied after debridement
  Ease-of-use as judged by attending physician on a VAS scale of 0=extremely difficult to use to 10=Very easy to use
Incidence of hematoma | At all treatments appointments until 3 weeks after STSG
  Nr of wounds which develop a hematoma
Inflammatory profiling of wound punch biopsies as assessed by mass spectrometry | Before STSG, 2 and 3 weeks and 12 months after STSG
  Mass spectrometry analysis of punch wound biopsies, investigating known inflammatory markers (TNF-alpha, IL-1b, IL-6, IL-8)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W. Shupp, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Burn Center at Medstar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided